CLINICAL TRIAL: NCT00499941
Title: Alpha-1 Foundation Research Registry
Status: Completed | Type: Observational
Sponsor: Medical University of South Carolina (Other)
Collaborators: Alpha-1 Foundation (Other)
Responsible Party: Principal Investigator, Charlie Strange, Professor of Pulmonary and Critical Care Medicine, Medical University of South Carolina
Other Study IDs: HR 9059
Record Dates: First submitted 2007-07-11; First posted 2007-07-12 (Estimated); Last update posted 2021-03-03 (Actual); Status verified 2021-02

CONDITIONS: Alpha 1-Antitrypsin Deficiency
Keywords: Alpha 1-Antitrypsin Deficiency
MeSH Terms: conditions — alpha 1-Antitrypsin Deficiency

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 20 Years
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The Alpha-1 Foundation Research Registry is a confidential database made up of individuals diagnosed with severe alpha-1 antitrypsin deficiency (Alpha-1) or the carrier state.

DETAILED DESCRIPTION:
The Registry was established in 1997 by the Alpha-1 Foundation to facilitate research initiatives and promote the development of improved treatments and a cure for Alpha-1. Located at the Medical University of South Carolina (MUSC) in Charleston, the Registry employs procedures that ensure the most stringent confidentiality of participants. The Registry operates under the direction of the Alpha-1 Foundation Board of Directors and is guided by an Advisory Committee comprised of leaders in the medical, ethical, scientific and Alpha communities. Individuals enrolled in the Registry have the ongoing opportunity to participate directly in clinical trials of new therapeutic approaches in addition to other research opportunities.

ELIGIBILITY:
Inclusion Criteria:

* Individuals of all ages who are diagnosed with severe alpha-1 antitrypsin deficiency or the carrier state

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Individuals of all ages who are diagnosed with severe alpha-1 antitrypsin deficiency or the carrier state
Sampling Method: Probability Sample
Enrollment: 6655 (Actual)
Dates: Start 2000-04; Primary Completion 2021-01 (Actual); Study Completion 2021-01 (Actual)

PRIMARY OUTCOMES:
To study the natural history of PiZZ, PiSZ, and PiMZ alpha-1 antitrypsin deficiency | Not limited

CONTACTS AND LOCATIONS:
Overall Officials: Charlie Strange, M.D., Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina. Division of Pulmonary and Critical Care Medicine, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Data sharing is encouraged by coordinator contact at MUSC

REFERENCES:
- [Background] Williams PH, Shore L, Sineath M, Quill J, Warner B, Keith J, Walker D, Wienke S, Flavin S, Strange C. Genetics' influence on patient experiences with a rare chronic disorder: a photovoice study of living with alpha-1 antitrypsin deficiency. Nurs Clin North Am. 2013 Dec;48(4):627-36. doi: 10.1016/j.cnur.2013.09.008. PMID 24295190
- [Background] Smith RA, Wienke S, Coffman DL. Alpha-1 couples: interpersonal and intrapersonal predictors of spousal communication and stress. J Genet Couns. 2014 Apr;23(2):212-20. doi: 10.1007/s10897-013-9639-6. Epub 2013 Aug 11. PMID 23934327
- [Background] Smith RA, Wienke SE, Baker MK. Classifying married adults diagnosed with alpha-1 antitrypsin deficiency based on spousal communication patterns using latent class analysis: insights for intervention. J Genet Couns. 2014 Jun;23(3):299-310. doi: 10.1007/s10897-013-9661-8. Epub 2013 Nov 1. PMID 24177906
- [Background] Holm KE, Wamboldt FS, Ford DW, Sandhaus RA, Strand M, Strange C, Hoth KF. The prospective association of perceived criticism with dyspnea in chronic lung disease. J Psychosom Res. 2013 May;74(5):450-3. doi: 10.1016/j.jpsychores.2013.02.001. Epub 2013 Feb 28. PMID 23597335
- [Background] Holm KE, Borson S, Sandhaus RA, Ford DW, Strange C, Bowler RP, Make BJ, Wamboldt FS. Differences in adjustment between individuals with alpha-1 antitrypsin deficiency (AATD)-associated COPD and non-AATD COPD. COPD. 2013 Apr;10(2):226-34. doi: 10.3109/15412555.2012.719049. PMID 23547634
- [Background] Hoth KF, Wamboldt FS, Strand M, Ford DW, Sandhaus RA, Strange C, Bekelman DB, Holm KE. Prospective impact of illness uncertainty on outcomes in chronic lung disease. Health Psychol. 2013 Nov;32(11):1170-4. doi: 10.1037/a0032721. Epub 2013 Jun 17. PMID 23772888
- [Background] Hoth KF, Ford DW, Sandhaus RA, Strange C, Wamboldt FS, Holm KE. Alcohol use predicts ER visits in individuals with alpha-1 antitrypsin deficiency (AATD) associated COPD. COPD. 2012 Aug;9(4):417-25. doi: 10.3109/15412555.2012.684414. Epub 2012 May 31. PMID 22651849
- [Result] Stoller JK, Brantly M, Fleming LE, Bean JA, Walsh J. Formation and current results of a patient-organized registry for alpha(1)-antitrypsin deficiency. Chest. 2000 Sep;118(3):843-8. doi: 10.1378/chest.118.3.843. PMID 10988213
- [Result] Bowlus CL, Willner I, Zern MA, Reuben A, Chen P, Holladay B, Xie L, Woolson RF, Strange C. Factors associated with advanced liver disease in adults with alpha1-antitrypsin deficiency. Clin Gastroenterol Hepatol. 2005 Apr;3(4):390-6. doi: 10.1016/s1542-3565(05)00082-0. PMID 15822045
- [Result] Eden E, Strange C, Holladay B, Xie L. Asthma and allergy in alpha-1 antitrypsin deficiency. Respir Med. 2006 Aug;100(8):1384-91. doi: 10.1016/j.rmed.2005.11.017. Epub 2006 Jan 5. PMID 16403617
- [Result] McGee D, Strange C, McClure R, Schwarz L, Erven M. The Alpha-1 Association Genetic Counseling Program: an innovative approach to service. J Genet Couns. 2011 Aug;20(4):330-6. doi: 10.1007/s10897-011-9355-z. Epub 2011 Mar 19. PMID 21424325
- See also: Alpha-1 Foundation Research Registry Website — http://www.alphaoneregistry.org